CLINICAL TRIAL: NCT01258283
Title: PET / CT With 18F-FDG (18F-fluorodeoxyglucose Positron Emission Tomography/Computed Tomography): Does it Optimize the I 123-MIBG (Iodine 123 Metaiodobenzylguanidine) Imaging Results in the Search for Discriminating Factors for the Implementation of an Implantable Defibrillator for Primary Prevention in Patients With Heart Failure of Ischemic Origin?
Brief Title: PET / CT With 18F-FDG: Does it Optimize the I 123-MIBG Imaging Results in the Search for Discriminating Factors for the Implementation of an Implantable Defibrillator?
Status: Terminated | Type: Observational
Why Stopped: Inclusion rate too slow / infeasible.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-I/2008/VB-03; 2008-007163-16 (Other: RCB number)
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2015-10

CONDITIONS: Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: See inclusion and exclusion criteria.
  Interventions: Other: Addional imaging

INTERVENTIONS:
Other: Addional imaging — All patients will systematically have an 18F-FDG PET-CT (18F-fluorodeoxyglucose positron emission tomography/computed tomography) and a 123MIBG (Iodine 123 metaiodobenzylguanidine) scintigraphy

SUMMARY:
The main objective of this study is to determine among the patients included a subpopulation that does not need a defibrillator.

This will be done by comparing the number of discordant segments (mismatch) between patients who have a severe arrhythmia (ventricular tachycardia or ventricular fibrillation) with appropriate electrical therapy within 3 years of monitoring and others. "Mismatch" in the definition of this objective is the usual definition: score 3.4 in I123-MIBG (Iodine 123 metaiodobenzylguanidine) and PET at 0,1,2.

ELIGIBILITY:
Inclusion Criteria:

* Patient with ischemic heart disease with heart failure
* Patients who received myocardial perfusion scintigraphy
* Indication for the implantation of an ICD installed according to current recommendations : LVEF <30% and NYHA (New York Heart Association) stage II, III.
* The subject must have given his informed consent and signed consent
* The subject must be a member or beneficiary of a social security system

Exclusion Criteria:

* Pregnant or lactating women
* History of "open heart" cardiovascular surgery
* Inability to sign informed consent (patient under guardianship)
* Patients with diabetes mellitus
* Patient with proven dementia
* Person refusing to sign the consent
* Someone who already has an ICD at baseline
* Life expectancy less than one year (NYHA IV, other diseases such as neoplastic disease in an advanced stage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary patients that should benefit from ICD (Implanted Cardiac Defibrillator) implantation for primary prevention according to current recommendations, that is to say with LVEF (left ventricular ejection fraction) <30% in NYHA (New York Heart Association) stage II or III and within one month of an myocardial infarction or within 3 months of a complete revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-06; Primary Completion 2015-08 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Presence/absence of a triggering of the defibrillator within 3 years of follow up | 3 years
  The primary endpoint is the triggering of the defibrillator within 3 years of follow up. Mismatch segments will be studied as predictors of arrhythmia.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Boudousq, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - Centre Hospitalier Universitaire de Montpellier, Montpellier